CLINICAL TRIAL: NCT04695210
Title: A Virtual Peer-to-peer Support Programme for Family Caregivers of Individuals with Motor Neurone Disease At Risk of Becoming or Currently Technology-dependent: Randomised Controlled Trial
Brief Title: Virtual Peer-to-peer Support Programme for Carers of MND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: MND Association (Unknown); Marie Curie Charity (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Louise Rose, Professor of Critical Care Nursing, King's College London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 292922
Record Dates: First submitted 2020-12-19; First posted 2021-01-05 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Motor Neuron Disease; Amyotrophic Lateral Sclerosis
Keywords: caregiver
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Parallel group single blinded (outcome assessor) randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Peer-to-Peer Support (Experimental): Those participants randomised to the intervention arm will have access to a 12-week virtual peer-to-peer support programme which entails:
  1. weekly audio, video, or text private messaging with a peer supporter;
  2. synchronous weekly discussion forum attended by peer supporters and family caregiver participants moderated by the research team. These forums will discuss specific topics (e.g. caregiver self-care, the emotional impact of caregiving). Ask the expert forums will be moderated by clinical experts every 6 weeks (meaning all participants will have access to 2 ask the expert sessions);
  3. asynchronous discussion forums in which participants can post questions; and
  4. access to informational resources.
  Interventions: Behavioral: Virtual peer-to-peer support
- Control (No Intervention): Those participants randomised to the control arm will receive usual care which comprises self-directed access to the MND Association Visitors programme and MND Association educational resources via their website.

INTERVENTIONS:
Behavioral: Virtual peer-to-peer support — See arm description
  Arms: Virtual Peer-to-Peer Support

SUMMARY:
Background/scope There is growing recognition that family caregiving is a serious public health issue requiring supportive interventions. Family caregivers play an essential role in sustaining a stable environment enabling individuals with motor neurone disease (MND) that are technology dependent to live at home. The family caregivers can experi¬ence exceptional burden and significant decline in psychological wellbeing due to MND's rapid and pro¬gressive nature with profoundly debilitating effects and intensive support needs. Dependence on assistive technology adds an additional level of complexity to family caregiving due to the need to learn how to operate and troubleshoot medical devices, train other caregivers, and negotiate appointments with new specialties within the healthcare system.

Despite the recognized impact of caregiving for individuals with MND, data are scarce as to effective interventions that provide direct practical and psychosocial supports. Difficulty accessing support may increase psychological distress. As the burden of caring increases due to disease progression and increasing technology dependence, access to existing informal support networks may diminish. Online peer support using virtual modalities is a flexible and low cost form of support. Peers, people who have experienced the same health problem and have similar characteristics as support recipients, can be a key source of emotional, informational, and affirmational support. Peer support improves psychological well-being of caregivers of people with conditions such as dementia, cancer, and brain injury. Although peer support programmes for family caregivers of people with MND exist, data as to their efficacy are limited. Therefore, we have developed an online peer support programme, completed beta and usability testing and now propose to test the effect on caregiver psychological wellbeing and caregiver burden.

Aim/research question(s) Overall aim: to determine the efficacy of a 12-week online peer support programme on family caregiver psychological health and caregiver burden.

Primary research question:

What is the effect of the online peer support programme on psychological distress measured using the Hospital Anxiety and Depression Scale (HADS)?

Secondary research questions:

1. What is the effect on positive affect, caregiver burden, caregiving mastery, caregiving personal gain, and coping?
2. How do participants use the programme (fidelity and reach)?
3. What is the perceived usability and acceptability?

Methods The investigators will conduct a parallel group randomised controlled trial with participants allocated to 12-week access to the online peer support programme or a usual care control group. The investigators will enrol family caregivers of an individual with MND who is referred for consideration or receiving any of the following

1. assisted ventilation
2. cough assist
3. gastroscopy and enteral feeding

i.e., entering King's clinical staging Stage 4A: nutritional support; or Stage 4B: respiratory support [51]:

The 12-week peer-to-peer support programme entails:

1. audio, video, or text private messaging;
2. synchronous weekly chat;
3. asynchronous discussion forum; and
4. informational resources.

The investigators will collect demographic and caregiving data including the Caregiver Assistance Scale and Caregiving Impact Scale, and caregiver measures (HADS, Positive and Negative Affect Schedule, Zarit Burden Interview, Pearlin Mastery Scale, Personal Gain Scale, Brief COPE) at baseline and programme completion.

The investigators will download use of online peer support programme features, assess usability, and conduct semi-structured interviews to explore acceptability using the Theoretical Framework of Acceptability.

To test for a medium size effect (d=0.5), at 5% level of significance (2-sided) with power 80%, 64 participants are required in each arm (128 total). Adjusting for 20% attrition requires 154 participants.

Proposed findings The proposed study will demonstrate the effect of a online peer support programme on psychological distress, positive affect, caregiving burden, mastery, personal gain and coping. Data on programme fidelity will enable the investigators to objectively assess acceptability and interpret study results. Data on usability and acceptability will inform future scalability of the online peer support programme outside of the trial both nationally and internationally, and to other family caregiver populations.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. family/informal caregiver of an individual with MND living at home who is referred for consideration or receiving any of the following i.e., entering King's clinical staging Stage 4A: nutritional support; or Stage 4B: respiratory support [51]:

   1. assisted ventilation
   2. cough assist
   3. gastroscopy and enteral feeding
3. able to speak/read English;
4. has access to a computer, tablet, or smartphone and the internet (we have the ability to provide loan 4G enabled tablets if required); and
5. consents to participation

Exclusion Criteria:

1. Actively receiving psychiatric/psychologist care identified through self-report.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Score (HADS) | 6 weeks & 12 weeks
  Change in Hospital Anxiety and Depression Score from baseline to programme completion. The Hospital Anxiety and Depression Score Overall score ranges from 0 [best] to 21 [worst] with cutoff points of >7 (possible) and >10 (probable) indicating cases of anxiety or depression.

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule | 12 weeks
  10-item Positive Affect Scale of the Positive and Negative Affect Schedule from baseline to programme completion. Scores range from 10 to 50; higher scores indicate more psychological well-being.
Zarit Burden Interview (ZBI) | 6 weeks & 12 weeks
  Change in ZBI score from baseline to programme completion. The sum of scores ranges between 0 to 88. Higher scores indicate greater burden. Caregivers can be categorised as 'highly burdened' (score of ≥ 24) and low burdened groups (score <24)
Pearlin Mastery Scale | 12 weeks
  Change in Pearlin Mastery Scale from baseline to programme completion. The Pearlin Mastery Scale is a 7 item scale with scores from 7 to 28. Higher scores indicate a greater sense of control over life.
Brief-COPE (note COPE is not an abbreviation) | 12 weeks
  Change in Brief COPE from baseline to programme completion. 14 scales with 2 items (28 items in total. Scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilisation of that specific coping strategy.

OTHER OUTCOMES:
Usability | At 12 weeks following programme completion
  For those participants in the intervention arm, on programme completion we will also ask them to rate the usability of the virtual peer-to-peer support programme on a 9-point Likert scale ranging from difficult to easy.
Acceptability | After 12 weeks following programme completion
  Semi-structured qualitative interviews exploring perceived acceptability of the virtual peer-to-peer support programme following programme completion

CONTACTS AND LOCATIONS:
Overall Officials: Louise Rose, PhD, Principal Investigator — King's College London
Locations (25):
- United Kingdom (25):
  - Bedfordshire Hospitals NHS Foundation Trust, Bedford
  - Airedale NHS Foundation Trust, Bradford
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - Pilgrims Hospice, Canterbury
  - Coventry Community Specialist Palliative Care Team, Coventry
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Ninewells Hospital, Dundee
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Phyllis Tuckwell Hospice, Farnham
  - Medway Community Healthcare, Gillingham
  - Kingston Hospital NHS Foundation, Kingston upon Thames
  - The Leicestershire & Rutland Organisation for the Relief of Suffering - LOROS, Leicester
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Lancashire Teaching Hospitals NHS Foundation Trust, Many Locations
  - Marie Curie Hospice, Many Locations
  - Nottinghamshire Healthcare NHS Foundation Trust, Many Locations
  - Swansea Bay University Health Board, Many Locations
  - Royal Stoke University Hospital/University Hospitals North, Multiple Locations
  - University Hospitals Plymouth NHS trust, Plymouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Severn Hospice, Shrewsbury
  - St Margaret's Hospice, Taunton
  - Hounslow and Richmond Community Healthcare, Teddington
  - Compton Care, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rose L, Thaventhiran T, Hobson E, Rogers R, James K, Chu P, Carter B, Faull C, Saha S, Lee JS, Kaltsakas G, McDermott C, Ramsay M. Digital peer-to-peer support programme for informal caregivers of people living with motor neuron disease: study protocol for a multi-centre parallel group, single-blinded (outcome assessor) randomised controlled superiority trial. Trials. 2023 Feb 20;24(1):119. doi: 10.1186/s13063-023-07124-3. PMID 36805758